CLINICAL TRIAL: NCT05740046
Title: Influence of Motor Intervention With the Intorus Tool on the Psychomotor Development of Children With Down Syndrome
Brief Title: Motor Intervention Whit the Intorus Tool on Children With Down Syndrome
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Extremadura (Other)
Responsible Party: Principal Investigator, Blanca González Sanchez, DOCTOR, University of Extremadura
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: ISD2023
Record Dates: First submitted 2023-01-30; First posted 2023-02-22 (Actual); Last update posted 2023-12-01 (Actual); Status verified 2023-11

CONDITIONS: Down Syndrome
Keywords: Down syndrome; psychomotoricity
MeSH Terms: conditions — Down Syndrome

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- experimental group (Experimental): Group that will receive the intervention sessions using the Intorus tool
  Interventions: Device: INTORUS
- control group (No Intervention): Group that will receive the intervention sessions without using the Intorus tool

INTERVENTIONS:
Device: INTORUS — INTERVENTION PROTOCOL WITH INTORUS
  Arms: experimental group

SUMMARY:
The goal of this clinical trial is to test in people with down syndrome how does the INTORUS tool influence their psychomotor development. The main question it aims to answer is:

- Does the INTORUS tool improve psychomotor development in people with Down Syndrome? The intervention program will be carried out during the Functional Habilitation sessions and will be carried out by the center's professionals. These sessions must be carried out in a quiet environment, without distractions so that the user can concentrate on carrying out the activities. It is important that the user attends the sessions in comfortable, sleeveless clothing, to allow the tool to slide smoothly through their upper limbs.

Each session will consist of several exercises with their corresponding rest breaks described in the Intervention Protocol. Each session attendance will be recorded following an attendance record model created for the occasion.

Participants will be divided into two groups randomly. The control group will receive an intervention treatment at the psychomotor level in the traditional way, following the protocols established in the center, and the intervention group will receive an intervention treatment at the psychomotor level with the INTORUS device.

Randomization will be carried out using the Oxford Minimization and Randomization software.

DETAILED DESCRIPTION:
POPULATION The population of interest are users of the Functional Habilitation Service of the Centers of the Down Syndrome Association of Cáceres and Plasencia

INCLUSION CRITERIA

* Users with Down Syndrome
* Ages between 4 and 18 years.
* Informed consent signed by parents/guardians.

EXCLUSION CRITERIA

* Users without Down Syndrome.
* Under 4 years and over 18 years.

A total of approximately 100 users will participate in the study. Participants will be divided into two groups randomly. The control group will receive an intervention treatment at the psychomotor level in the traditional way, following the protocols established in the center, and the intervention group will receive an intervention treatment at the psychomotor level with the INTORUS device.

Randomization will be carried out using the OxMaR (Oxford Minimization and Randomization) software.

PROJECT REGISTRATION The project has been approved by the Bioethics and Biosafety Commission of the University of Extremadura as of 12/19/2022.

INTERVENTION PROGRAM

The intervention program will be carried out during the Functional Habilitation sessions and will be carried out by the center's professionals. These sessions must be carried out in a quiet environment, without distractions so that the user can concentrate on carrying out the activities. It is important that the user attends the sessions in comfortable, sleeveless clothing, to allow the tool to slide smoothly through their upper limbs.

Each session will consist of several exercises with their corresponding rest breaks described in the Intervention Protocol. Each session attendance will be recorded following an attendance record model created for the occasion.

INTERVENTION PROTOCOL

To carry out the intervention sessions, all participants will follow the same protocol for the use of INTORUS. It is a protocol created for the study of increasing difficulty in which the participants advance to a higher level once they have passed the lower level.

EVALUATION

The evaluations will be carried out prior to the start of treatment, at 20 weeks of treatment and at 40 weeks of treatment once the intervention program has concluded.

The tools used to carry out the evaluation will be:

* Questionnaire of participating sociodemographic variables
* Pediatric Balanced Scale (PBS)
* Berg Balance Scale
* Harris test. Adaptation of the Harris Test of Lateral Dominance
* Single leg support time on a stable surface
* Satisfaction questionnaire for professionals
* Participant satisfaction questionnaire adapted to easy reading. The evaluations will be carried out by a professional external to the treatment to avoid bias.

Once the intervention period is over, a questionnaire will be passed to the professionals participating in the study to assess the usefulness of the device, the degree of satisfaction with it and the usefulness of the therapies applied, and a satisfaction questionnaire for participants adapted for easy reading. to know the degree of satisfaction and usefulness of the tool on the part of the participants.

TIMELINE

The intervention consists of 40 treatment sessions lasting 45 minutes each with a frequency of 2 days a week in which the intervention protocol described in Annex 7 described above will be developed. (15 min from Intorus) Previously, the participants will receive a "session 0" in which they will carry out a first contact with the device.

ELIGIBILITY:
Inclusion Criteria:

* Users with Down Syndrome
* Ages between 4 and 18 years.
* Informed consent signed by parents/guardians.

Exclusion Criteria:

* Users without Down Syndrome.
* Under 4 years and over 18 years

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 30 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2023-07-31 (Actual)

PRIMARY OUTCOMES:
Change in Pediatric Balanced Scale | Before starting the interventions, at 3 months and at 6 months at the end of the study.
  The Pediatric Balance Scale is a modified version of the Berg Balance Scale that is used to assess functional balance skills in school-aged children. The scale consists of 14 items that are scored from 0 points (lowest function) to 4 points (highest function) with a maximum score of 56 points
Change in Berg Equilibrium Scale | Before starting the interventions, at 3 months and at 6 months at the end of the study.
  Scale for measuring balance in people over 15 years of age. The Berg Balance Scale (BBS) is used to objectively determine a patient's ability (or inability) to safely balance during a series of predetermined tasks. It is a 14 item list with each item consisting of a five-point ordinal scale ranging from 0 to 4, with 0 indicating the lowest level of function and 4 the highest level of function and takes approximately 20 minutes to complete. It does not include the assessment of gait.

SECONDARY OUTCOMES:
Change in Harris test | Before starting the interventions, at 3 months and at 6 months at the end of the study.
  Scale for assessing lateralisation. In this way, it is possible to find out whether the child has a rightward, leftward, ambidextrous, incomplete, crossed or opposite laterality dominance.

OTHER OUTCOMES:
PROFESSIONAL SATISFACTION | through study completion, an average of 5 months
  Questionnaire to measure the degree of satisfaction of the professionals participating in the study with the use of the tool.
PARTICIPANTS SATISFACTION | through study completion, an average of 5 months
  Questionnaire to measure the degree of satisfaction of the participants in the study with the use of the tool.

CONTACTS AND LOCATIONS:
Overall Officials: BLANCA GONZÁLEZ SÁNCHEZ, DOCTOR, Principal Investigator — UNIERSIDAD DE EXTREMADURA
Locations (1):
- Blanca Gonzalez Sanchez, Cáceres, Spain

IPD SHARING:
Plan to Share IPD: No